CLINICAL TRIAL: NCT00004902
Title: Phase II Pilot Evaluation of Infusional 8 Cl-cAMP in the Treatment of Relapsed or Refractory Multiple Myeloma
Brief Title: Tocladesine in Treating Patients With Recurrent or Refractory Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: NU FDA97H4; NU-97H4; NCI-G00-1681
Record Dates: First submitted 2000-03-07; First posted 2004-07-26 (Estimated); Last update posted 2012-05-30 (Estimated); Status verified 2012-05

CONDITIONS: Multiple Myeloma and Plasma Cell Neoplasm
Keywords: refractory multiple myeloma; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — 8-chloro-cyclic adenosine monophosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: tocladesine

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of tocladesine in treating patients who have recurrent or refractory multiple myeloma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the safety of 8-chloro-cyclic adenosine monophosphate (8-chloro-cAMP) in patients with recurrent or refractory multiple myeloma. II. Evaluate the efficacy of this regimen in these patients. III. Determine the pharmacokinetics of this regimen in these patients.

OUTLINE: Patients receive 8-chloro-cyclic adenosine monophosphate (8-chloro-cAMP) over 120 hours every 2 weeks for up to 4 courses. Beginning with course 5, patients with stable or responsive disease receive 8-chloro-cAMP over 120 hours every 3 weeks until disease progression. Patients are followed every 3 months until death.

PROJECTED ACCRUAL: A maximum of 29 patients will be accrued for this study within 12-18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed recurrent or refractory multiple myeloma Measurable disease by monoclonal serum or urine globulins OR Malignant plasma cells documented on bilateral bone marrow biopsy Refractory after at least one prior therapeutic regimen (no more than 2 prior regimens allowed)

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: Creatinine no greater than 1.5 mg/dL AND/OR Creatinine clearance at least 60 mL/min Calcium no greater than 8.7 g/dL Cardiovascular: No history of arrhythmias No uncontrolled angina pectoris No symptomatic coronary ischemia No grade 3 or 4 congestive heart failure Cardiac ejection fraction greater than 35% by gated imaging Other: Not pregnant or nursing Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: At least 3 weeks since prior chemotherapy Endocrine therapy: At least 3 weeks since prior glucocorticoids Radiotherapy: Not specified Surgery: Not specified Other: No concurrent theophylline therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1998-01; Primary Completion 1999-11 (Actual); Study Completion 1999-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ann Traynor, MD, Study Chair — Robert H. Lurie Cancer Center
Locations (1):
- Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois, United States